CLINICAL TRIAL: NCT00000353
Title: Efficacy/Safety Trial of Buprenorphine/Nx for Opiate Dependence
Brief Title: Trial of Buprenorphine/Naloxone for Opiate Dependence - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-2; Y01-3-0012-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a buprenorphine/naloxone sublingual tablet formulation as an office-based therapy for opiate dependence treatment.

ELIGIBILITY:
Please contact site for information.

Ages: 19 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-10; Primary Completion 1997-09 (Actual); Study Completion 1997-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States